CLINICAL TRIAL: NCT03854006
Title: Cryoballoon Pulmonary Vein Isolation: Time-to-Isolation Dependent Freeze Protocols Comparison
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Izabela Warchol, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22012019
Record Dates: First submitted 2019-02-16; First posted 2019-02-26 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The investigators will examine long-term efficacy of Cryo-AF using the two proposed dosing algorithms in a nonrandomized fashion.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze cycle: 240 s - TTI <75 s or 2x240 s - >75 s (Active Comparator): In the first group freeze duration is 240s if TTI (time-to-isolation) is < 75 s. In case of TTI>75s a 240s bonus freeze is applied.
  If no TTI could be documented, a single 240 s freeze cycle is applied in this group in case of balloon temperature -40°C (degrees Celsius) after 60 s.
  Interventions: Procedure: Cryoballoon pulmonary vein isolation
- Freeze cycle: TTI+120 s (Active Comparator): In the second group freeze duration is TTI (time-to-isolation) +120 s. If no TTI could be documented, a single 180 s freeze cycle is applied in this group in case of balloon temperature -40 °C after 60 s.
  Interventions: Procedure: Cryoballoon pulmonary vein isolation

INTERVENTIONS:
Procedure: Cryoballoon pulmonary vein isolation — During cryoballoon pulmonary vein isolation, under local anaesthesia, diagnostic catheters are placed in the coronary sinus. The cryoballoon is advanced to the left atrium via a steerable sheath after single transseptal puncture and inflated at the PV(pulmonary vein) ostia. A spiral mapping catheter is advanced through the balloon inner lumen and positioned in the PV at the closest achievable proximity to the cryoballoon in order to record real-time PV potentials during PV isolation. During PV isolation the potentials from the PV are recorded. The TTI is defined as the time of the last recording of a PV potential before sustained isolation. Isolation of all PVs is reassessed at the end of the procedure by documentation of entrance- and exit-block.

SUMMARY:
The purpose of this study is to develop and prospectively test two Cryo-AF (atrial fibrillation) dosing protocols guided exclusively by time-to-isolation (TT-I) in patients undergoing a first-time Cryo-AF.

Both protocols guided by TT-I are associated with shorter cryoapplications as compared to conventional approach.

In the first group freeze duration is TTI +120 s. In the second group freeze duration is 240s if TTI is < 75 s. In case of TTI>75s a 240s bonus freeze is applied.

The investigators examine long-term efficacy of Cryo-AF using the two proposed dosing algorithms in a nonrandomized fashion.

The study cohort consists of consecutive patients undergoing a first-time Cryo-AF for symptomatic paroxysmal or persistent AF (atrial fibrillation) at Interventional Cadiology and Cardiac Arrhythmias Clinic of Medical University in Łódź. During 12 months investigators are planning to enroll 40 patients Patients are randomly assigned to the groups. All of them will be followed up 3 and 12 months after the procedure. In addition, ambulatory electrocardiographic monitoring will also be performed at 3 and 12 months.

The study is requested for an approval of the university ethics committee.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Paroxysmal or Persistent Atrial Fibrillation on Electrocardiogram

Exclusion Criteria:

Diagnosis of Sinus Rhythm on Electrocardiogram

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation Recurrence | 3 months after the procedure
Atrial Fibrillation Recurrence | 12 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Lubinski, MD, PhD, Study Director — Medical University of Lodz
Locations (1):
- Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej - Centralny Szpital Weteranów, Lodz, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided